CLINICAL TRIAL: NCT02115984
Title: Double-blind Multicenter Placebo-controlled Study of the Safety and Leukostimulatory Activity of the Preparation "Panagen" in Patients With Breast Cancer
Brief Title: Study of the Safety and Leukostimulatory Activity of the Preparation "Panagen" in Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Panagen, Limited Liability Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-bc-2
Record Dates: First submitted 2014-04-07; First posted 2014-04-16 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy & Panagen (Experimental): Panagen 5 mg tablet by mouth every 2-3 h (six times a day) for 18 days. Patients start to receive the preparation immediately after the chemotherapy and take three tablets during 6 h, that is one tablet every 2 h. Then the patients stop taking the preparation and resume its administration after 42 h, that is, 48 h after the chemotherapy (Day 3) and continue its administration for 17 days (to Day 20 after the chemotherapy).
  Interventions: Drug: Panagen; Procedure: Chemotherapy
- Chemotherapy & Placebo (Placebo Comparator): Placebo tablet by mouth every 2-3 h (six times a day) for 18 days. Patients start to receive the placebo tablets immediately after the chemotherapy and take three tablets during 6 h, that is one tablet every 2 h. Then the patients stop taking the preparation and resume its administration after 42 h, that is, 48 h after the chemotherapy (Day 3) and continue its administration for 17 days (to Day 20 after the chemotherapy).
  Interventions: Drug: Placebo; Procedure: Chemotherapy

INTERVENTIONS:
Drug: Panagen
  Other Names: sodium deoxyribonucleate; double-stranded human DNA
  Arms: Chemotherapy & Panagen
Drug: Placebo
  Arms: Chemotherapy & Placebo
Procedure: Chemotherapy — Chemotherapy course includes 500 mg/m2 cyclophosphan, 50 mg/m2 doxorubicin, and 500 mg/m2 fluorouracil administered intravenously in one day.

SUMMARY:
The goal of this trial is to assess the safety, therapeutic dose, and leukostimulatory activity of the preparation Panagen in the therapeutic schemes for treating cancer diseases in the patients receiving a standard chemotherapy for breast cancer of stages II-IV (with distant metastases).

DETAILED DESCRIPTION:
The limited liability company Panagen has designed the preparation named Panagen in a form of tablets, which is represented by a fragmented nucleoprotein complex isolated from the human placenta. The method allows for extraction of a full-fledged genomic DNA with retention of its fragments that are tightly associated with the nuclear matrix proteins. The length of fragmented DNA varies from 200 to 6000 base pairs.

This trial is a double-blind multisite placebo-controlled sequentially randomized phase II trial involving two groups of patients. Totally, 80 stage II breast cancer cases with an increased risk or stage III-IV breast cancer cases (with distant metastases) requiring chemotherapy will participate in this trial. All patients will be sequentially randomized, that is, any patient independently of the time she is included into this study may fall into one of the two groups. The patients will be divided into two groups at a ratio of 3 : 1; the first group receiving the preparation Panagen will contain 60 persons and the second one, receiving placebo, 20 persons. For the reasons of ethics, the size of the second group minimally possible for obtaining statistically significant data is chosen. The patients will be subject to a standard chemotherapy, including 500 mg/m2 cyclophosphan, 50 mg/m2 doxorubicin, and 500 mg/m2 fluorouracil; all preparations are administered intravenously once a day. In this trial, the patients will receive three chemotherapy courses with an interval of 3 weeks between the courses (unless an interruption is required).

On the background of this chemotherapy, the patients will receive the preparation Panagen at a dose of 30 mg/day or a placebo with a fractional uniform administration during the active day period, which will amount to one tablet six times a day (every 2 h). The patients start to receive the preparation immediately after the chemotherapy and take three tablets during 6 h, that is one tablet every 2 h. Then the patients stop taking the preparation and resume its administration after 42 h, that is, 48 h after the chemotherapy (day 3) and continue its administration for 17 days to and thorough day 20 after the chemotherapy. If the next chemotherapy course is delayed, the patients continue taking Panagen. The intake should be stopped 1 day before the next chemotherapy course. It is admissible to delay the next chemotherapy course by 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Women at an age of ≥18 years
* Stage II-IV breast cancer (with distant metastases)
* The patients will be subject to chemotherapy with cyclophosphan/doxorubicin/ fluorouracil as a standard chemotherapy for treating breast cancer
* The patients have not been earlier subject to chemotherapy
* Functional status according to the Eastern Cooperative Oncology Group (ECOG) ≤2
* Leukocyte counts of ≥3 × 109/L before the treatment course
* Neutrophil counts of ≥1.5 × 109/L before the treatment course
* Platelet counts of ≥100 × 109/L before the treatment course
* Adequate heart function
* Adequate liver function, that is, alanine aminotransferase / aspartate aminotransferase (ALT / AST) activity < 2.5 × upper limit of normal (ULN); acid phosphatase activity < 5 × ULN; and bilirubin concentration < 5 × ULN; and
* Adequate renal function, that is, the creatinine concentration in the blood serum < 1.5 × ULN; urea concentration < ULN; and endogenous creatinine clearance

Exclusion Criteria:

* Participation in clinical trials less than 30 days before sequential randomization
* Previous exposure to Panagen or any other leukostimulatory drugs at a stage of clinical development
* Known hypersensitivity to cyclophosphan, doxorubicin, or fluorouracil
* Therapy with systemically active antibiotics less than 72 h before the beginning of chemotherapy
* Long-term oral intake of corticosteroids
* Previous X-ray therapy performed less than 4 weeks before randomization
* Previous transplantation of hematopoietic stem cells
* Other malignant neoplasms during the last 5 years except for basal cell or flat cell carcinoma or intraepithelial carcinoma of the uterine cervix
* Any disease or state that according to the opinion of researcher can influence patient's safety or the estimation of a final trial point; and
* Pregnant and nursing women; the fertile patients should use chemical or barrier contraceptives during the period of trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

REFERENCES:
- [Derived] Proskurina AS, Gvozdeva TS, Potter EA, Dolgova EV, Orishchenko KE, Nikolin VP, Popova NA, Sidorov SV, Chernykh ER, Ostanin AA, Leplina OY, Dvornichenko VV, Ponomarenko DM, Soldatova GS, Varaksin NA, Ryabicheva TG, Uchakin PN, Rogachev VA, Shurdov MA, Bogachev SS. Five-year disease-free survival among stage II-IV breast cancer patients receiving FAC and AC chemotherapy in phase II clinical trials of Panagen. BMC Cancer. 2016 Aug 18;16:651. doi: 10.1186/s12885-016-2711-5. PMID 27538465
- [Derived] Proskurina AS, Gvozdeva TS, Alyamkina EA, Dolgova EV, Orishchenko KE, Nikolin VP, Popova NA, Sidorov SV, Chernykh ER, Ostanin AA, Leplina OY, Dvornichenko VV, Ponomarenko DM, Soldatova GS, Varaksin NA, Ryabicheva TG, Uchakin PN, Zagrebelniy SN, Rogachev VA, Bogachev SS, Shurdov MA. Results of multicenter double-blind placebo-controlled phase II clinical trial of Panagen preparation to evaluate its leukostimulatory activity and formation of the adaptive immune response in patients with stage II-IV breast cancer. BMC Cancer. 2015 Mar 13;15:122. doi: 10.1186/s12885-015-1142-z. PMID 25886605

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy & Panagen | Chemotherapy & Placebo
Started | 57 | 23
Completed | 51 | 16
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy & Panagen | Chemotherapy & Placebo | Total
Number analyzed (Participants) | 57 | 23 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (7) | 53 (8) | 52 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 23 | 80
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Quantity of Leukocytes and Neutrophils in the Blood of Patients
Time Frame: Baseline, Day 21 after 2nd chemotherapy (Day 42 post-baseline), Day 21 after 3rd chemotherapy (Day 63 post-baseline)
Measure: Median (Inter-Quartile Range); unit: 10^9 cells/L
Arm/Group | Chemotherapy & Panagen | Chemotherapy & Placebo
Number analyzed (Participants) | 51 | 16
10^9 cells/L
  Leukocytes baseline | 8.1 [6.5 to 8.8] | 7.2 [6.5 to 7.9]
  Leukocytes after the 2nd chemotherapy | 6.6 [5.9 to 7.2] | 4.8 [4.1 to 5.6]
  Leukocytes after the 3rd chemotherapy | 5 [4.6 to 5.5] | 4.1 [3.8 to 4.4]
  Neutrophils baseline | 5.33 [4.42 to 6.36] | 5.2 [4.2 to 6.05]
  Neutrophils after the 2nd chemotherapy | 4.62 [3.43 to 4.82] | 2.76 [2.22 to 3.27]
  Neutrophils after the 3rd chemotherapy | 3.19 [1.81 to 3.58] | 2.44 [2.31 to 2.63]

ADVERSE EVENTS:
Description: Some Serious Adverse Events and Other (Not Including Serious) Adverse Events were estimated not for all patients, but only for 33 from Panagen group and 11 from Placebo group.
Arm/Group | Chemotherapy & Panagen | Chemotherapy & Placebo
Serious Adverse Events (participants affected / at risk) | 57/57 | 23/23
Other Adverse Events (participants affected / at risk) | 1/33 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Chemotherapy & Panagen (N=57) | Chemotherapy & Placebo (N=23)
Herpetic eruption (Immune system disorders) | 0/33 | 3/11
Dry skin (Skin and subcutaneous tissue disorders) | 15/33 | 9/11
Dry eyes (Eye disorders) | 13/33 | 2/11
Heartburn (Gastrointestinal disorders) | 9/33 | 2/11
Alopecia (Skin and subcutaneous tissue disorders) | 57 | 23
Nausea after the CT (before day 7) (Gastrointestinal disorders) | 57 | 23
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy & Panagen (N=33) | Chemotherapy & Placebo (N=11)
Flatulence (Gastrointestinal disorders) | 1 | 0
Hive-like allergic reaction (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No